CLINICAL TRIAL: NCT03180255
Title: Multi-Center, Double-Masked, Randomized, Placebo-Controlled Phase 2b Clinical Trial Designed to Evaluate the Safety and Efficacy of Iontophoretic Dexamethasone Phosphate Ophthalmic Solution in Patients Having Undergone Cataract Surgery With Implantation of a Posterior Chamber Intraocular Lens (IOL)
Brief Title: Iontophoretic Delivery of EGP-437 in Patients Who Have Undergone Cataract Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eyegate Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGP-437-009
Record Dates: First submitted 2017-06-05; First posted 2017-06-08 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Cataract; Anterior Chamber Inflammation; Pain, Postoperative
MeSH Terms: conditions — Cataract; Pain, Postoperative | interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Intervention Model Description: Double-masked, randomized, placebo-controlled, multi-center, Phase 2b clinical trial designed to evaluate the efficacy and safety of transcleral iontophoretic delivery of dexamethasone phosphate ophthalmic solution in patients having undergone cataract surgery with implantation of a monofocal posterior chamber IOL.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor, investigator, subject will all be masked to study treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EGP-437 (Experimental): 40 mg/ml dexamethasone phosphate solution delivered by iontophoresis treatment consisting of 4.5 mA-min at 3.0 mA
  Interventions: Combination Product: Dexamethasone phosphate
- Placebo (Placebo Comparator): 100 mM sodium citrate buffer solution (placebo) delivered by iontophoresis treatment consisting of 4.5 mA-min at 3.0 mA
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: Dexamethasone phosphate — Ocular iontophoretic delivery of a steroid
  Arms: EGP-437
Other: Placebo — Ocular iontophoretic delivery of a placebo
  Other Names: Sodium Citrate Buffer
  Arms: Placebo

SUMMARY:
Phase 2b trial evaluating the safety and efficacy of EGP-437, versus placebo using the EyeGate® II Drug Delivery System (EGDS) in patients having undergone cataract surgery with implantation of a monofocal posterior chamber intraocular lens (IOL).

DETAILED DESCRIPTION:
This will be a Phase 2b, double-masked, multi-site study, in which a total of up to 100 eyes of up to 100 subject will be enrolled at up to 8 clinical sites in the United States. The study has 2 different treatment arms consisting of the following iontophoresis treatment regimen:

Treatment Arm 1, up to 50 subjects will receive the following study treatment:

40 mg/ml dexamethasone phosphate solution delivered by iontophoresis treatment consisting of 4.5 mA-min at 3.0 mA on Day 0 (immediately following cataract surgery), Day 1 (24 hours' post-cataract surgery), Day 4, and a potential Day 7 treatment that will be administered for subjects who have ≥11 AC cells per high-power field on slit lamp examination.

Treatment Arm 2, up to 50 subjects will receive the following study treatment:

100 mM sodium citrate buffer solution (placebo) delivered by iontophoresis treatment consisting of 4.5 mA-min at 3.0 mA on Day 0 (immediately following cataract surgery), Day 1 (24 hours' post-cataract surgery), Day 4, and a potential Day 7 treatment that will be administered for subjects who have ≥11 AC cells per high-power field on slit lamp examination.

Subjects will come in for 6 visits over 28 days.

The primary efficacy endpoint (PEP) will evaluate 1) the proportion of subjects with an AC cell count of zero on Day 7 and 2) the proportion of subjects with a pain score of zero on Day 1.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing unilateral cataract extraction and implantation of a monofocal IOL (at the time of enrollment)
2. Age 18 to 85 years
3. Receive, understand, and sign a copy of the written informed consent form (ICF)
4. Are able to return for all study visits and willing to comply with all study-related instructions

Exclusion Criteria:

1. Are undergoing implantation of a multifocal and/or depth enhancing IOL
2. Are undergoing or have just undergone cataract surgery on the study eye that is deemed complex or may require manipulation of the iris
3. The study eye has a small pupil or iris requiring manipulation due to synechiae and/ Tamsulosin (Flomax®, Boehringer Ingelheim) use
4. Have a Seidel positive wound following surgical procedure despite suture and/or ReSure® Sealant placement
5. Have had ocular surgery of any kind in the study eye within 3 months prior to baseline visit (Day 0)
6. Have undergone cataract surgery in the fellow eye within 4 weeks prior to baseline visit (Day 0) and still require post-operative medications in that fellow eye
7. Are scheduled for surgery in the fellow eye within the study period
8. Have anterior chamber inflammation as measured by slit lamp examination in the study eye at the baseline visit (Day 0) [Defined as anterior chamber (AC) cell and/or flare grade > 0]
9. Have history of uveitis or inflammatory disease in the study eye
10. Requires simultaneous supplemental surgery, such as glaucoma procedures or vitrectomy, in the study eye
11. Have used any topical ocular medication in either eye, other than tear substitute for dry eye, within the past 2 weeks prior to baseline visit (Day 0)
12. Have used topical corticosteroid or nonsteroidal anti-inflammatory drug (NSAID) treatment in either eye < 48 hours prior to the baseline visit (Day 0) (excluding the use of topical NSAIDs, pre-operatively on Day 0 and administered at the clinic site under the investigator's oversight)
13. Have IOP ≥ 25 mmHg at baseline, a history of glaucoma, and/or require ocular anti-hypertensive medications
14. Are known corticosteroid IOP responder in study eye
15. Have received systemic administration of corticosteroid and/or immunosuppressants within the past 14 days prior to baseline visit (Day 0)
16. Have received intravitreal, sub-Tenon, or any periocular corticosteroid treatment in either eye within the past 6 months prior to baseline visit (Day 0)
17. Have open wounds/skin disease on the forehead area where the iontophoresis return electrode will be applied
18. Have lesions of the eyelids or the ocular surface impeding the application of the iontophoresis applicator
19. Have blepharospasm, blepharophimosis, or other eyelid anatomic variations precluding placement of the iontophoresis applicator
20. Have known allergy to dexamethasone or dexamethasone phosphate or any medication to be used in this study
21. Have history or diagnosis of ocular herpes, corneal lesion of suspected herpetic origin that could be worsened with steroid use
22. Have optic neuritis of any origin
23. Have clinically suspected or confirmed central nervous system or ocular lymphoma
24. Have active hyphema, pars planitis, choroiditis, toxoplasmosis scar, vitreous hemorrhage, and/or clinically significant macular edema (CSME) that would compromise visual acuity recovery
25. Have severe/serious ocular pathology or medical condition which may preclude study completion
26. Have pacemaker and/or any other electrical sensitive support system
27. Are pregnant or lactating female, or female of childbearing age and using inadequate birth control method
28. Have participated in another investigational device or drug study within 30 days of baseline visit (Day 0) (other clinical trial participation while participating in EGP-437-009 would be prohibited per protocol)
29. Have previously participated in a study with EGP-437

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
AC cell count = 0 | 7 days' following first study treatment
  The proportion of subjects with an AC cell count of zero on Day 7
Pain score = 0 | 1 day post-surgery and following first study treatment
  The proportion of subjects with a pain score of zero on Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brandano, BS, Study Director — VP, Clinical Operations
Locations (1):
- Site 901, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No